CLINICAL TRIAL: NCT00006182
Title: Stroke Prevention in Sickle Cell Anemia (STOP 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 68; U01HL052016 (NIH)
Record Dates: First submitted 2000-08-21; First posted 2000-08-22 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-10

CONDITIONS: Blood Disease; Cerebrovascular Accident; Anemia, Sickle Cell
MeSH Terms: conditions — Hematologic Diseases; Stroke; Anemia, Sickle Cell | interventions — Blood Transfusion

INTERVENTIONS:
Procedure: Blood Transfusion

SUMMARY:
To determine how long blood transfusions are needed for primary stroke prevention. Also, to determine the duration of risk associated with abnormal transcranial Doppler ultrasound (TCD) and to determine the specificity of the stroke risk model developed in STOP 1 in patients with abnormal TCD measurements.

DETAILED DESCRIPTION:
BACKGROUND:

Without intervention, 11 percent of children with sickle cell anemia will sustain a stroke before the age of 20. The STOP 2 follows on the recently completed NHLBI trial, Stroke Prevention Trial in Sickle Cell Anemia (STOP 1), which found that patients at high risk for stroke could be identified using transcranial Doppler (TCD) ultrasound, and that the incidence of stroke could be reduced by 90 percent in those children by periodic blood transfusion for at least 36 months. However, chronic intermittent blood transfusions are cumbersome, expensive and associated with morbidity from iron overload. Thus, this study to determine if transfusion can be safely halted after 30 months of treatment is critically important to the continued clinical care of patients with sickle cell disease at risk for stroke.

DESIGN NARRATIVE:

In this multicenter, randomized clinical trial, 100 children will be randomized to continue to receive periodic transfusion therapy and 50 to discontinue receiving periodic transfusion therapy. The primary endpoint will be the reversion of the transcranial Doppler velocity levels to greater than 200 cm/second, indicating return of increased risk for overt stroke. Recruitment will be in two phases. Phase I will include those patients who began transfusions before April 1, 1999. These will come mainly from the STOP 1 cohort. Those who begin transfusions after April 1, 1999 but before April 1, 2001 will be eligible for Phase II of recruitment. All patients will receive quarterly TCD examinations. Patients who revert to high risk will be offered return to transfusion. The overall design includes a three month start-up, the two phases of recruitment (established STOP patients and new patients) for a total of 36 months, 18 months of observations after recruitment ends and then 3 months of wrap-up.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-07; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Adams — Augusta University; Donald Brambilla — New England Research Institutes, Inc.

REFERENCES:
- [Background] Vichinsky EP, Luban NL, Wright E, Olivieri N, Driscoll C, Pegelow CH, Adams RJ; Stroke Prevention Trail in Sickle Cell Anemia. Prospective RBC phenotype matching in a stroke-prevention trial in sickle cell anemia: a multicenter transfusion trial. Transfusion. 2001 Sep;41(9):1086-92. doi: 10.1046/j.1537-2995.2001.41091086.x. PMID 11552063
- [Background] Kral MC, Brown RT. Transcranial Doppler ultrasonography and executive dysfunction in children with sickle cell disease. J Pediatr Psychol. 2004 Apr-May;29(3):185-95. doi: 10.1093/jpepsy/jsh020. PMID 15131136
- [Background] Wang WC, Morales KH, Scher CD, Styles L, Olivieri N, Adams R, Brambilla D; STOP Investigators. Effect of long-term transfusion on growth in children with sickle cell anemia: results of the STOP trial. J Pediatr. 2005 Aug;147(2):244-7. doi: 10.1016/j.jpeds.2005.02.030. PMID 16126058
- [Result] Adams RJ, Brambilla D; Optimizing Primary Stroke Prevention in Sickle Cell Anemia (STOP 2) Trial Investigators. Discontinuing prophylactic transfusions used to prevent stroke in sickle cell disease. N Engl J Med. 2005 Dec 29;353(26):2769-78. doi: 10.1056/NEJMoa050460. PMID 16382063
- [Derived] Adamkiewicz TV, Abboud MR, Paley C, Olivieri N, Kirby-Allen M, Vichinsky E, Casella JF, Alvarez OA, Barredo JC, Lee MT, Iyer RV, Kutlar A, McKie KM, McKie V, Odo N, Gee B, Kwiatkowski JL, Woods GM, Coates T, Wang W, Adams RJ. Serum ferritin level changes in children with sickle cell disease on chronic blood transfusion are nonlinear and are associated with iron load and liver injury. Blood. 2009 Nov 19;114(21):4632-8. doi: 10.1182/blood-2009-02-203323. Epub 2009 Aug 31. PMID 19721013